CLINICAL TRIAL: NCT00812656
Title: Serial Measurement of a Plasma Stroke Biomarker Panel in Patients Undergoing Cardiac Surgery With Cardiopulmonary Bypass
Acronym: Stroke08
Status: Completed | Type: Observational
Sponsor: Klinikum Ludwigshafen (Other)
Responsible Party: Prof. Dr. J. Boldt, Klinikum Ludwigshafen
Other Study IDs: StrokePanel08
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stroke Panel group: Patients undergoing cardiac surgery with the use of cardiopulmonary bypass

SUMMARY:
The purpose of this study is to investigate changes in new plasma stroke biomarker panel in patients undergoing cardiac surgery with the use of cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Elective cardiac surgery with the use of cardiopulmonary bypass

Exclusion Criteria:

* Patients undergoing emergent procedures
* Patients with preoperative mechanical support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac surgery with the use of cardiopulmonary bypass
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in stroke index | day before surgery; first and second day postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Stefan W Suttner, MD, Principal Investigator — Klinikum Ludwigshafen
Locations (1):
- Klinikum Ludwigshafen, Ludwigshafen, RLP, Germany